CLINICAL TRIAL: NCT05182983
Title: Tongue Image Database and Diagnostic Model for Digestive Tract Disease Diagnosis
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Gang Chen, MD, Clinical Professor, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Other Study IDs: Gasinthep tongue image
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Digestive Tract Diseases; Liver Diseases; Colorectal Disease; Gastric Diseases; Small Bowel Disease
MeSH Terms: conditions — Liver Diseases; Stomach Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with digestive tract diseases
  Interventions: Other: Tongue images，coating on the tongue and clinical data
- Healthy people
  Interventions: Other: Tongue images，coating on the tongue and clinical data

INTERVENTIONS:
Other: Tongue images，coating on the tongue and clinical data — Take photos of the tongue of patients with gastrointestinal diseases and collect clinical information.

SUMMARY:
The tongue images of patients with gastrointestinal diseases and healthy people will be collected and the tongue image database will be established. Through deep learning and artificial intelligence, early screening models of various gastrointestinal tumors based on tongue images were constructed.

ELIGIBILITY:
Inclusion Criteria:

1. Be older than 18 years old;
2. Clinical or pathological diagnosis of Digestive tract diseases;
3. Patients before receiving surgery, chemotherapy, radiotherapy, targeted therapy, local therapy, immunotherapy and other treatment measures；
4. The patient had no tongue disease
5. Patients understand and are willing to sign written informed consent.

Exclusion Criteria:

1. Patients unable to complete the process as required (mental disorder or poor compliance, etc.);
2. The patient or guardian is unwilling to participate in this study;
3. Combined with other serious systemic diseases (heart failure, renal failure,hematopoietic system disease or Uncontrollable acute infection);

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with gastrointestinal diseases and healthy people
Sampling Method: Non-Probability Sample
Enrollment: 10690 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Diagnosis | 1 year
  The differences of tongue images between patients with digestive tract diseases and healthy people

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, M.D., Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- Gang Chen, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No